CLINICAL TRIAL: NCT00001858
Title: Monitoring for Donor-Specific Hyporesponsiveness Following Renal and Pancreatic Allotransplantation
Brief Title: Monitoring for Tolerance to Kidney or Combined Kidney-Pancreas Transplants
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990119; 99-DK-0119
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-05-30

CONDITIONS: Graft Rejection; Kidney Disease
Keywords: Biopsy; Immune System; Renal
MeSH Terms: conditions — Kidney Diseases

SUMMARY:
This protocol facilitates the development of methods for determining whether transplant recipients have developed immune hyporesponsiveness or tolerance towards their allograft. These methods will involve the study of peripheral blood or biopsy tissue obtained at regular intervals from patients receiving kidney or combined kidney-pancreas allografts at the Warren G. Magnuson Clinical Center. In addition, patients that have previously received a kidney or combined kidney-pancreas allograft will be evaluated using assays requiring peripheral blood mononuclear cells and/or biopsies. Assays developed under this protocol will be used in subsequent protocols to assess the effects of immune modulating treatment regimens and may eventually be used to direct clinical care or guide the withdrawal of immunosuppressive agents. However, patients enrolled in this protocol will not have any change in treatment based solely on the assays developed without being enrolled in an additional study.

DETAILED DESCRIPTION:
This protocol facilitates the development of methods for determining whether transplant recipients have developed immune hyporesponsiveness or tolerance towards their allograft. These methods will involve the study of peripheral blood or biopsy tissue obtained at regular intervals from patients receiving kidney or combined kidney-pancreas allografts at the Warren G. Magnuson Clinical Center. In addition, patients that have previously received a kidney or combined kidney-pancreas allograft will be evaluated using assays requiring peripheral blood mononuclear cells and/or biopsies. Assays developed under this protocol will be used in subsequent protocols to assess the effects of immune modulating treatment regimens and may eventually be used to direct clinical care or guide the withdrawal of immunosuppressive agents. However, patients enrolled in this protocol will not have any change in treatment based solely on the assays developed without being enrolled in an additional study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney or combined kidney-pancreas transplant performed at the National Institutes of Health, or non-uremic healthy volunteers who are not on immunosuppressive medications.

Previous recipients of kidney or combined kidney-pancreas transplants.

Recipients of kidney or combined kidney-pancreas transplants interested in participation in the Recurrent Disease Allograft Registry.

Willingness and legal ability to give informed consent or permission from a legal guardian.

Willingness to travel to the Clinical Center for protocol specific samples to be taken, or in some cases, the ability to send samples via overnight mail.

For transplant patients, availability of donor tissue for testing. This could include splenic or peripheral blood lymphocytes from a cadaveric donor or a willing living donor enrolled on the Clinical Center Living Donor Protocol who consents to periodic phlebotomy for peripheral blood lymphocyte isolation.

EXCLUSION CRITERIA:

Inability or unwillingness to comply with protocol monitoring and therapy, including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services, or access to anti-rejection drugs after the research protocol is completed.

Any active malignancy. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing these are appropriately eliminated prior to transplant.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol allograft biopsies.

Platelet count less than 100,000/mm(3).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 1999-06-08; Study Completion 2014-05-30

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Matas AJ, Gillingham KJ, Sutherland DE. Half-life and risk factors for kidney transplant outcome--importance of death with function. Transplantation. 1993 Apr;55(4):757-61. doi: 10.1097/00007890-199304000-00014. PMID 8475549
- [Background] Najarian JS, Chavers BM, McHugh LE, Matas AJ. 20 years or more of follow-up of living kidney donors. Lancet. 1992 Oct 3;340(8823):807-10. doi: 10.1016/0140-6736(92)92683-7. PMID 1357243
- [Background] Santiago-Delpin EA. Trends in kidney transplantation in the United States. Transplant Proc. 1998 Sep;30(6):2867-8. doi: 10.1016/s0041-1345(98)00846-x. No abstract available. PMID 9745602